CLINICAL TRIAL: NCT04053569
Title: Effects of Polyphenols From a Table Grape on the Lipidomic Profile and Serum LDL Fractions: Possible Implications in the Metabolic Syndrome
Brief Title: Grape Polyphenols and Metabolic Syndrome
Acronym: PolyGrape
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Francesco Russo, Director of Nutritional Pathophysiology Laboratory - IRCCS S. de Bellis, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC2019019
Record Dates: First submitted 2019-08-06; First posted 2019-08-12 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Syndrome, Protection Against
Keywords: polyphenols; diet; lipidomics; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind clinical trial
Who Masked: Participant
Masking Description: Single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet with table grape (Experimental): Table grape (5g/Kg) administered for four weeks with dietary recommendations. A strict restriction of fruits and the limitation of other foods containing polyphenols will be necessary.
  Interventions: Dietary Supplement: Table Grape supplement
- Specific dietary advice (No Intervention): Dietary recommendations (such as limitation of alcohol, caffeine), and low consumption of fruits.

INTERVENTIONS:
Dietary Supplement: Table Grape supplement — 5g/Kg of table grape for four weeks with dietary recommendations along with a strict restriction of fruits and limitation of other foods containing polyphenols.
  Arms: Diet with table grape

SUMMARY:
Fruits and vegetables are beneficial for patients with metabolic syndrome, a condition characterized by the coexistence of various risk factors (obesity, hypertension, hypercholesterolemia, insulin resistance) that predispose to cardiovascular disease and diabetes. Diets such as the Mediterranean diet, rich in flavonoids and polyphenolic compounds can exert a high anti-inflammatory, antithrombotic and antiproliferative action. Several studies have shown that grape polyphenols exert a crucial protective action against the onset of cardiovascular, neurodegenerative, and cancer diseases. On the other hand, little information is available on the health effects deriving from the consumption of table grapes on cell membranes lipidomic profile. On this basis, the aim of this study is the evaluation of possible changes in lipidomic profile and plasma antioxidant activity induced by a diet enriched with table grape polyphenols.

DETAILED DESCRIPTION:
Purified polyphenols extracted by table grape can decrease cell proliferation in vitro and exert anti-atherosclerotic and antithrombotic activities, regulating endothelial function. Literature studies have already evaluated the cytostatic and apoptotic effects produced by table grape extracts from different cultivars, demonstrating a different behavior based on extract composition. The beneficial effects of polyphenols have been attributed exclusively to their direct antioxidant action; however, in recent years it has emerged that polyphenols can interact with intracellular signaling mechanisms, modulating the activity of transcription factors involved in cell lipid metabolism. Lipidomic analysis studies the lipids in a "dynamic" way, monitoring the changes in membrane phospholipids content, caused by inflammation, stress, or malnutrition. These changes can also affect the cellular and plasmatic prothrombotic potential, which results altered in metabolic diseases. Recently, alterations in erythrocytes lipidomic profile have been detected in subjects with steatosis. Moreover, in patients with colorectal cancer patients, the presence of metastases at the time of surgery was associated with an altered profile of fatty acids in the membrane of colonic tissue cells.

Moreover, data in literature show how diet and functional foods can modify serum lipid content, in particular, an important role in the onset of dysmetabolic diseases is undoubtedly played by the different fractions of Low-Density Lipoproteins (LDL). The presence of smaller LDL fractions in the serum, such as fraction 3 and fraction 4, has been associated with the onset of cardiovascular disease and myocardial infarctions. Therefore, understanding the molecular mechanisms underlying the effects of nutraceuticals is essential to develop prevention and intervention strategies on subjects at risk for metabolic syndrome.

On this basis, the aim of this study is the evaluation of possible changes happening in lipidomic profile, plasma antioxidant activity and plasma prothrombotic potential induced by a diet enriched with table grape polyphenols in subjects with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age > 30 years and <65 years
* overweight.

Exclusion Criteria:

* cardiovascular disease.
* stroke
* treatment with insulin or oral hypoglycemic drugs
* fasting glucose > 126 mg / dl, or casual glycemia > 200 mg / dl
* more than 20 g/day of alcohol intake
* serious medical conditions that may compromise participation in the trial
* subjects following a special diet or involved in a weight-loss program or unable to follow a diet for religious or other reasons.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in serum concentrations (mg/dL) of cholesterol, triglycerides, glucose | Before the start of the study (time 0), after four weeks (time 1) and after eight weeks (time 2)
  Blood samples will be taken after at least 12 hours of fasting and the concentrations of cholesterol. triglycerides, and glucose will be assessed according to the standard laboratory methods (commercially available kits).
Changes in blood concentration of fatty acids (stearic acid, oleic acid, arachidonic acid, eicosaepentanoic acid) expressed as percentage (%) | Before the start of the study (time 0) and after eight weeks (time 2)
  All human blood samples are treated with chloroform: methanol (2:1, v/v), and the samples are centrifuged. The lower layer, containing fatty acids, are removed with care, replaced in a new tube and dried by a centrifugal evaporator. The fatty acid methyl ester (FAME) is obtained by adding toluene and BF3. Samples are collected and transferred into a vial and analyzed by gas chromatography.
Changes in serum concentration of single subfractions of LDL (expressed as mg/dL) | Before the start of the study (time 0) and after eight weeks (time 2)
  Small dense LDL analysis: Small dense Lipoproteins (sdLDL) are assayed using Lipoprint LDL System (Quantimetrix, USA). Each serum sample is applied on high resolution polyacrylamide gel tube in order to separate LDL fractions and subfractions by electrophoresis. The resolved lipoproteins bands are scanned and analyzed.

SECONDARY OUTCOMES:
Changes in the concentrations of radical monocation of 2,2'-azinobis-(3-ethylbenzothiazoline-6-sulfonic acid) (ABTS) expressed as µM Trolox equivalents/g of dry weight | Before the start of the study (time 0), after four weeks (time 1) and after eight weeks (time 2)
  The ABTS assay will be performed using the commercially available ZENBIO-AOX-1 kit.
Changes in plasma prothrombotic potential | Before the start of the study (time 0), after four weeks (time 1) and after eight weeks (time 2)
  The plasma prothrombotic potential will be evaluated using a functional test able to monitor the entire kinetics of thrombin generation, including its inactivation by plasma physiological inhibitors. In these tests, the coagulation will be activated by purified tissue factor.
Changes in plasma grape miRNA content | Before the start of the study (time 0) (time 1) and after eight weeks (time 2)
  Total serum RNA, including Small RNAs, will be extracted from plasma (200µL) of the subjects involved in the study using the miRNeasy Mini Kit (QIAGEN). After checking the concentration and quality, the effective presence of miRNAs will be verified by retro-transcription with a specific miRNA kit (TaqMan miRNA Reverse Transcription kit - Life Technologies) using Real Time-polymerase chain reaction (PCR) method.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Notarnicola, ScD, Principal Investigator — IRCCS "Saverio de Bellis" Castellana Grotte
Locations (1):
- IRCCS Saverio de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li B, Zhang C, Zhan YT. Nonalcoholic Fatty Liver Disease Cirrhosis: A Review of Its Epidemiology, Risk Factors, Clinical Presentation, Diagnosis, Management, and Prognosis. Can J Gastroenterol Hepatol. 2018 Jul 2;2018:2784537. doi: 10.1155/2018/2784537. eCollection 2018. PMID 30065915
- [Background] Liu YC, Chen WL, Kung WH, Huang HD. Plant miRNAs found in human circulating system provide evidences of cross kingdom RNAi. BMC Genomics. 2017 Mar 14;18(Suppl 2):112. doi: 10.1186/s12864-017-3502-3. PMID 28361700
- [Background] Mlotshwa S, Pruss GJ, MacArthur JL, Endres MW, Davis C, Hofseth LJ, Pena MM, Vance V. A novel chemopreventive strategy based on therapeutic microRNAs produced in plants. Cell Res. 2015 Apr;25(4):521-4. doi: 10.1038/cr.2015.25. Epub 2015 Feb 27. No abstract available. PMID 25721325
- [Background] Notarnicola M, Caruso MG, Tutino V, Bonfiglio C, Cozzolongo R, Giannuzzi V, De Nunzio V, De Leonardis G, Abbrescia DI, Franco I, Intini V, Mirizzi A, Osella AR. Significant decrease of saturation index in erythrocytes membrane from subjects with non-alcoholic fatty liver disease (NAFLD). Lipids Health Dis. 2017 Aug 23;16(1):160. doi: 10.1186/s12944-017-0552-0. PMID 28830448
- [Background] Ammollo CT, Semeraro F, Milella RA, Antonacci D, Semeraro N, Colucci M. Grape intake reduces thrombin generation and enhances plasma fibrinolysis. Potential role of circulating procoagulant microparticles. J Nutr Biochem. 2017 Dec;50:66-73. doi: 10.1016/j.jnutbio.2017.08.012. Epub 2017 Sep 1. PMID 29040837